CLINICAL TRIAL: NCT02720172
Title: A Randomized Trial of an Early Postoperative Home Exercise Program Versus Usual Care After Anterior Cervical Discectomy and Fusion Surgery
Brief Title: Early Postoperative Home Exercise Program After Cervical Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Kristin Archer, Associate Professor and Vice Chair of Research, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150912
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Spinal Fusion; Cervical Spine Degenerative Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Home Exercise Program (Experimental): The early home exercise program is an exercise-based self-management program for patients immediately after cervical spine surgery.
  Interventions: Behavioral: Early Home Exercise Program
- Usual Care (Other): Usual postoperative care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Early Home Exercise Program — The early home exercise program is a 6-week program of home exercises with weekly phone calls to monitor progression and compliance.
  Arms: Early Home Exercise Program
Other: Usual Care — Usual care involves standard postoperative management under the direction of the treating surgeon.
  Arms: Usual Care

SUMMARY:
The overall objective of this two-group randomized controlled trial is to gather preliminary evidence on the efficacy and safety of early postoperative exercise for improving disability, pain, and general physical health in patients after anterior cervical discectomy and fusion (ACDF) surgery. Our central hypothesis is that an early home exercise program (HEP) performed within the first six weeks after surgery will decrease disability and pain and improve general health, through increases in physical activity and self-efficacy and reductions in fear of movement. The results of our randomized trial will advance research on postoperative management for patients with cervical spine surgery and provide evidence in line with a value-based healthcare approach for optimizing outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Surgical treatment of a cervical degenerative condition (cervical stenosis, spondylosis, degenerative spondylolisthesis, disc herniation) using anterior cervical discectomy and fusion procedure;
2. English speaking due to feasibility of employing study personnel to deliver and assess the study intervention; and
3. Age older than 21 years (younger individuals do not typically have a cervical degenerative condition)

Exclusion Criteria:

1. Patients having surgery secondary to trauma, fracture, tumor, infection, or spinal deformity;
2. Patients undergoing cervical corpectomy;
3. Diagnosis or presence of severe psychiatric disorder such as schizophrenia or other psychotic disorder, including but not limited to Brief Psychotic disorder and Delusional disorder;
4. Documented history of alcohol and/or drug abuse;
5. Patients having surgery under a workman's compensation claim; and
6. Unable to provide a stable telephone or physical address

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | Up to 12 months after surgery
  The NDI measures disease-specific disability for cervical spine patients.
Numeric Rating Scale (NRS) | Up to 12 months after surgery
  The NRS measures levels of neck and arm pain intensity.
12-Item Short Form Health Survey (SF-12) | Up to 12 months after surgery
  The SF-12 is a measure of general physical and mental health.

SECONDARY OUTCOMES:
Movement Accelerometry | Up to 12 months after surgery
  Movement accelerometry measures general physical activity level.

OTHER OUTCOMES:
Fusion rate | 6 months after surgery
  Fusion rate will be measured using dynamic flexion-extension radiograph.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin R Archer, PhD, DPT, Principal Investigator — Vanderbilt University Medical Center; Rogelio A Coronado, PT, PhD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No